CLINICAL TRIAL: NCT06015334
Title: Applying Virtual Reality to Compare Visual Performance Following Bilateral Implantation of TECNIS Synergy vs TECNIS Monofocal Intraocular Lens With Monovision in Patients With Cataract: A Randomized Controlled Trial.
Brief Title: Assessment of Visual Performance With Virtual Reality After Cataract Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: The University of Hong Kong (Other)
Collaborators: Janssen, LP (Industry)
Responsible Party: Principal Investigator, Professor Christopher K.S. Leung, Clinical Professor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: H022_Protocol_VR Cataract
Record Dates: First submitted 2023-08-23; First posted 2023-08-29 (Actual); Last update posted 2023-08-29 (Actual); Status verified 2023-08

CONDITIONS: Cataract
Keywords: cataract; virtual reality; multifocal intraocular lens; trifocal intraocular lens; monovision
MeSH Terms: conditions — Cataract | interventions — Cataract Extraction; Lens Implantation, Intraocular

STUDY DESIGN:
Intervention Model Description: Patients with cataract will receive implantation of bilateral trifocal IOL (TECNIS Synergy) implantation or bilateral monofocal IOL (Tecnis monofocal) with monovision.
Who Masked: Participant
Masking Description: Patients will remain unaware of their specific study arm assignments until the completion of the study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Bilateral implantation of trifocal intraocular lens (Active Comparator): Patients will receive bilateral implantation of TECNIS Synergy intraocular lens
  Interventions: Procedure: cataract surgery with implantation of intraocular lens
- Bilateral monofocal intraocular lens implantation with monovision (Active Comparator): Patients will receive bilateral implantation of TECNIS monofocal intraocular lens
  Interventions: Procedure: cataract surgery with implantation of intraocular lens

INTERVENTIONS:
Procedure: cataract surgery with implantation of intraocular lens — Cataract surgery with implantation of bilateral trifocal IOL (TECNIS Synergy) implantation or bilateral monofocal IOL (Tecnis monofocal) with monovision.

SUMMARY:
The proposed randomized clinical trial aims to compare visual performance, measured using VR simulations, in cataract patients implanted either with bilateral trifocal IOL or bilateral monofocal IOL with monovision. The hypothesis is that patients implanted with trifocal IOL would exhibit superior visual performance, in both daytime and nighttime conditions, compared to those with a monofocal IOL with monovision.

DETAILED DESCRIPTION:
Cataract surgery provides an opportunity to restore the quality of life by improving vision. While monofocal intraocular lenses (IOLs) implantation with monovision has been a common approach for cataract surgery, it may result in limited clarity at the intermediate distance and reduced depth perception. The advent of multifocal IOLs has expanded the possibilities, potentially offering increased visual performance in different ranges of vision. However, the benefits of multifocal IOLs in everyday activities are not fully understood due to the lack of task-based investigations.

To address this gap, a virtual reality-based approach is proposed to simulate daily activities and assess visual performance. This innovative method can provide insights into how multifocal IOLs enhance activities requiring good binocular vision at varying distances, a capability monofocal IOLs may lack. A randomized clinical trial is suggested to compare the TECNIS Synergy multi-focal IOL with the TECNIS monofocal IOL in monovision. Unlike its bifocal predecessors, the TECNIS Synergy IOL is trifocal, providing clear vision at near, intermediate, and far distances. The hypothesis is that patients implanted with the TECNIS Synergy IOL will demonstrate superior visual performance in simulated day and night conditions compared to those implanted with monofocal IOLs and monovision.

ELIGIBILITY:
Inclusion Criteria:

* Bilateral cataract
* Regular corneal astigmatism
* Corneal endothelium cell count >2000 cells/mm2
* Clear intraocular media other than cataract

Exclusion Criteria:

* Concomitant ocular diseases
* Irregular corneal aberration
* Capsular instability
* Systemic disease that may affect vision
* History of other intraocular surgery

Min Age: 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 114 (Estimated)
Dates: Start 2023-10-01 (Estimated); Primary Completion 2024-09-30 (Estimated); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
Overall Virtual reality (VR) performance score | Pre-operation, Month3
  VR performance score measured from all VR simulations

SECONDARY OUTCOMES:
Task-specific VR performance score | Pre-operation, Month3
  VR performance score measured from an individual VR simulation
Binocular reading speed assessment | Pre-operation, Month3
  Reading speed assessed by the MNRead acuity chart
Binocular contrast sensitivity | Pre-operation, Month3
  Contrast sensitivity assessed by Pelli-Robson contrast sensitivity chart
Distance visual acuity | Pre-operation, Day1, Week1, Month1, Month3
  Monocular and binocular uncorrected and corrected distance visual acuity
Intermediate (66 cm) visual acuity | Month3
  Monocular and binocular uncorrected and distance-corrected intermediate (66 cm) visual acuity
Near (40 cm) visual acuity | Month3
  Monocular and binocular uncorrected and distance-corrected near (40 cm) visual acuity
Binocular defocus curve | Month3
  Binocular defocus curve (from +1.0D to -4.0D) under photopic conditions (85 candela [cd]/m2)
Photic phenomena | Pre-operation, Month3
  Evaluation of photic phenomena by the 30-item quality of vision questionnaire
Quality of life assessment | Pre-operation, Month3
  National Eye Institute 25-item Visual Function Questionnaire Rasch score

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Leung, MD, MB ChB, Principal Investigator — The University of Hong Kong

IPD SHARING:
Plan to Share IPD: No
Our plan is focused on publishing the analyzed results of our research through peer-review, journals and conference papers. We understand the importance of patient privacy and confidentiality. Therefore, we will not share any individual patient data with any third parties.

REFERENCES:
- [Background] Zhang F, Sugar A, Jacobsen G, Collins M. Visual function and spectacle independence after cataract surgery: bilateral diffractive multifocal intraocular lenses versus monovision pseudophakia. J Cataract Refract Surg. 2011 May;37(5):853-8. doi: 10.1016/j.jcrs.2010.12.041. PMID 21511153
- [Background] Mahrous A, Ciralsky JB, Lai EC. Revisiting monovision for presbyopia. Curr Opin Ophthalmol. 2018 Jul;29(4):313-317. doi: 10.1097/ICU.0000000000000487. PMID 29708928
- [Background] Chen M, Atebara NH, Chen TT. A comparison of a monofocal Acrysoft IOL using the "blended monovision" formula with the multifocal array IOL for glasses independence after cataract surgery. Ann Ophthalmol (Skokie). 2007 Fall;39(3):237-40. doi: 10.1007/s12009-007-0035-4. PMID 18025632
- [Background] Goldberg DG, Goldberg MH, Shah R, Meagher JN, Ailani H. Pseudophakic mini-monovision: high patient satisfaction, reduced spectacle dependence, and low cost. BMC Ophthalmol. 2018 Nov 9;18(1):293. doi: 10.1186/s12886-018-0963-3. PMID 30413145
- [Background] Smith CE, Allison RS, Wilkinson F, Wilcox LM. Monovision: Consequences for depth perception from large disparities. Exp Eye Res. 2019 Jun;183:62-67. doi: 10.1016/j.exer.2018.09.005. Epub 2018 Sep 17. PMID 30237103
- [Background] Lam AKN, To E, Weinreb RN, Yu M, Mak H, Lai G, Chiu V, Wu K, Zhang X, Cheng TPH, Guo PY, Leung CKS. Use of Virtual Reality Simulation to Identify Vision-Related Disability in Patients With Glaucoma. JAMA Ophthalmol. 2020 May 1;138(5):490-498. doi: 10.1001/jamaophthalmol.2020.0392. PMID 32191274
- [Background] Dick HB, Ang RE, Corbett D, Hoffmann P, Tetz M, Villarrubia A, Palomino C, Castillo-Gomez A, Tsai L, Thomas EK, Janakiraman P. Comparison of 3-month visual outcomes of a new multifocal intraocular lens vs a trifocal intraocular lens. J Cataract Refract Surg. 2022 Nov 1;48(11):1270-1276. doi: 10.1097/j.jcrs.0000000000000971. Epub 2022 May 12. PMID 35545816
- [Background] Ferreira TB, Ribeiro FJ, Silva D, Matos AC, Gaspar S, Almeida S. Comparison of refractive and visual outcomes of 3 presbyopia-correcting intraocular lenses. J Cataract Refract Surg. 2022 Mar 1;48(3):280-287. doi: 10.1097/j.jcrs.0000000000000743. PMID 34321410
- [Background] Ramulu PY, Swenor BK, Jefferys JL, Rubin GS. Description and validation of a test to evaluate sustained silent reading. Invest Ophthalmol Vis Sci. 2013 Jan 23;54(1):673-80. doi: 10.1167/iovs.12-10617. PMID 23258146
- [Background] Mangione CM, Lee PP, Gutierrez PR, Spritzer K, Berry S, Hays RD; National Eye Institute Visual Function Questionnaire Field Test Investigators. Development of the 25-item National Eye Institute Visual Function Questionnaire. Arch Ophthalmol. 2001 Jul;119(7):1050-8. doi: 10.1001/archopht.119.7.1050. PMID 11448327
- [Background] Mangione CM, Lee PP, Pitts J, Gutierrez P, Berry S, Hays RD. Psychometric properties of the National Eye Institute Visual Function Questionnaire (NEI-VFQ). NEI-VFQ Field Test Investigators. Arch Ophthalmol. 1998 Nov;116(11):1496-504. doi: 10.1001/archopht.116.11.1496. PMID 9823352
- [Background] Petrillo J, Cano SJ, McLeod LD, Coon CD. Using classical test theory, item response theory, and Rasch measurement theory to evaluate patient-reported outcome measures: a comparison of worked examples. Value Health. 2015 Jan;18(1):25-34. doi: 10.1016/j.jval.2014.10.005. PMID 25595231
- See also: Probabilistic Models for Some Intelligence and Attainment Tests — https://www.semanticscholar.org/paper/Probabilistic-Models-for-Some-Intelligence-and-Rasch/d3203958e1b9c007d06340aad11d41f088875f3e#citing-papers